CLINICAL TRIAL: NCT05959967
Title: The Efficacy of Vestibular Rehabilitation Exercises and General Fitness Training pn Dizziness, Balance Confidence, and Mobility in Individuals With Bilateral Vestibular Hypofunction: A Randomized Controlled Trial
Brief Title: Vestibular Rehabilitation Exercises vs. General Fitness Training on Dizziness, Balance Confidence, and Mobility in Individuals With Bilateral Vestibular Hypofunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VRGFT2023
Record Dates: First submitted 2023-07-18; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Vestibular Disorder
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two groups: the VRE group or the GFT group.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular Rehabilitation Exercises (VRE) (Experimental): The VRE arm will be engaged in vestibular exercises including gaze stabilization, balance, and gait training.
  Interventions: Behavioral: Vestibular Rehabilitation Exercises
- General Fitness Training (GFT) (Active Comparator): The GFT arm will participate in general fitness exercises including cardiovascular, strength, and flexibility training.
  Interventions: Behavioral: General Fitness Training

INTERVENTIONS:
Behavioral: Vestibular Rehabilitation Exercises — The VRE group will receive exercises aimed at improving gaze stability, postural control, and balance. This includes activities like gaze stabilization exercises, balance training on different surfaces, and walking with head movements.
  Arms: Vestibular Rehabilitation Exercises (VRE)
Behavioral: General Fitness Training — The GFT group will undertake exercises to enhance cardiovascular fitness, strength, and flexibility, such as light aerobic exercises, resistance training, and stretching. The exercise sessions will be 60 minutes in duration, consisting of a warm-up phase, the main exercise phase, and a cool-down phase.
  Arms: General Fitness Training (GFT)

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of Vestibular Rehabilitation Exercises (VRE) and General Fitness Training (GFT) in adults diagnosed with vestibular disorders. The main questions it aims to answer are:

Does VRE lead to better improvements in gaze stabilization, balance, and gait than GFT? Does GFT lead to more improvements in overall fitness than VRE? Participants will be randomly assigned to either the VRE or GFT group and will participate in 60-minute exercise sessions twice weekly for 8 weeks. Researchers will compare the improvements in the two groups to see which intervention is more effective.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18 - 60 years.
* Diagnosis of a vestibular disorder confirmed by a healthcare professional.
* Able to walk unassisted for at least 10 meters.
* Able to understand and comply with the procedures of this study.
* Willing to provide informed consent.

Exclusion Criteria:

* Severe cardiovascular, respiratory, or metabolic disease that contraindicates physical exercise.
* Neuromuscular disorders that may affect balance and mobility other than the diagnosed vestibular disorder.
* History of orthopedic surgery within the past 6 months.
* Currently participating in another interventional clinical trial.
* Pregnant or breastfeeding women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-25 (Estimated); Primary Completion 2024-02-25 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Vertigo Symptom Scale (VSS) Scores from Baseline to 8 Weeks | Changes between Baseline and 8 weeks
  This outcome is the difference in scores on the Vertigo Symptom Scale (VSS), a validated vestibular symptom questionnaire, from baseline to 8 weeks. The VSS has two components: a vertigo/balance scale, with a score range of 0-36, and an autonomic/anxiety scale, with a score range of 0-28. Higher scores on both scales indicate more severe symptoms.
Change in Biodex Balance System Scores from Baseline to 8 Weeks | Baseline and 8 weeks
  This outcome is the difference in scores on the Biodex Balance System, a validated tool for balance assessment, from baseline to 8 weeks. The Biodex Balance System assesses participants' ability to maintain postural control through a variety of tests, including the Stability Index, Fall Risk Test, and Postural Stability Test. Lower scores on the Stability Index indicate better balance, while lower scores on the Fall Risk and Postural Stability tests indicate lower risk of falling and better postural stability, respectively.

SECONDARY OUTCOMES:
Change in Six-Minute Walk Test (6MWT) Distance from Baseline to 8 Weeks | Baseline and 8 weeks
  This outcome is the difference in the distance covered during the Six-Minute Walk Test (6MWT) from baseline to 8 weeks. The 6MWT assesses the maximum distance that can be walked in 6 minutes. A greater distance indicates better cardiovascular fitness.
Change in Flexibility Test Scores from Baseline to 8 Weeks | Baseline and 8 weeks
  This outcome is the difference in scores on a standard flexibility test, such as the Sit and Reach Test, from baseline to 8 weeks. The test assesses the flexibility of the lower back and hamstring muscles. A greater reach distance or score indicates better flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No